CLINICAL TRIAL: NCT00008775
Title: Pressure Support Ventilation During CF Exacerbations: A Randomized, Controlled Trial
Brief Title: Pressure Support Ventilation During CF Exacerbations
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Cystic Fibrosis Foundation (Other)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NCRR-M01RR00400-0654
Record Dates: First submitted 2001-01-16; First posted 2001-01-18 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

INTERVENTIONS:
Device: Pressure support ventilation

SUMMARY:
Chest physiotherapy is recognized as a mainstay of cystic fibrosis therapy, and is particularly important during treatment of pulmonary exacerbations. For some patients, especially those with moderate to severe compromise of lung function, this therapy may impose a high demand in the work of breathing and energy expenditure. The goal of this study is to evaluate the effectiveness of adding pressure support ventilation (PSV) during chest physiotherapy sessions in patients with cystic fibrosis with moderate to severe lung function compromise being treated for a pulmonary exacerbation.

DETAILED DESCRIPTION:
The proposed study will be conducted over three years. Cystic fibrosis patients with moderate to severe pulmonary disease who are experiencing an acute exacerbation that requires hospitalization will be admitted to the GCRC. Subject participation in the study will be for the first 10 days of hospitalization. Subjects will be randomized into one of two treatment groups: usual care or usual care plus non-invasive pressure support ventilation (PSV).

ELIGIBILITY:
cystic fibrosis subjects with pulmonary exacerbation

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States